CLINICAL TRIAL: NCT02544308
Title: Phase III Randomised Trial of Immunomodulatory Therapy in High Risk Solitary Bone Plasmacytoma
Brief Title: Trial of Immunomodulatory Therapy in High Risk Solitary Bone Plasmacytoma
Acronym: IDRIS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/13/0291
Record Dates: First submitted 2015-07-28; First posted 2015-09-09 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Plasmacytoma
Keywords: Solitary, Bone
MeSH Terms: conditions — Plasmacytoma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No further treatment (Active Comparator): No further treatment
  Interventions: Other: No further treatment
- Lenalidomide + Dexamethasone (Experimental): Lenalidomide 25mg orally daily on days 1-21 Dexamethasone 20mg orally on days 1, 8, 15 & 22 Up to 9 cycles
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Experimental Arm
  Other Names: Revlimid
  Arms: Lenalidomide + Dexamethasone
Drug: Dexamethasone — Experimental Arm
  Arms: Lenalidomide + Dexamethasone
Other: No further treatment — Comparator Arm
  Arms: No further treatment

SUMMARY:
The purpose of the trial is to establish whether adjuvant therapy with lenalidomide + dexamethasone after radiotherapy can improve progression free survival in patients with high risk solitary bone plasmacytoma compared with RT only.

DETAILED DESCRIPTION:
Solitary bone plasmacytoma (SBP) is a localised proliferation of malignant plasma cells (PCs) in the skeleton. The annual UK incidence is 0.4/100,000 (lower than multiple myeloma (MM)) with a peak age incidence at 68 years and there are estimated to be about 260 new cases per year in the United Kingdom (UK). The majority of patients with SBP ultimately progress to myeloma and this is likely due to occult disease not detected by conventional staging methods. Standard care for these patients is involved field radiotherapy (IFRT), but despite radical doses, two-thirds develop multiple myeloma at a median of 2 years, more so if there are high risk features.

The IDRIS Trial is a phase III study where the investigators hope to demonstrate that adjuvant lenalidomide + dexamethasone following IFRT prevents the development of multiple myeloma in patients with high risk solitary bone plasmacytoma. Whilst a proportion of solitary bone plasmacytoma is cured with IFRT, it is clear that the majority will progress to multiple myeloma. The investigators are seeking to prevent this outcome by using adjuvant therapy in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly-diagnosed SBP
* SBP treated with local radiotherapy with curative intent (see appendix 2).
* Radiotherapy completed within 28 days of registration
* Age ≥18 years
* ECOG performance status 0-2
* Written informed consent
* Willing to comply with the requirements of the Celgene pregnancy prevention programme

Exclusion Criteria:

* Multifocal plasmacytoma, solitary extramedullary plasmacytoma or myeloma
* ≥10% bone marrow plasma cells
* Clinical suspicion of failure to respond to radiotherapy
* Receiving or intention to treat with systemic corticosteroid therapy (e.g. dexamethasone or prednisolone) unless otherwise agreed by the TMG
* Severe hepatic impairment (bilirubin >2xULN or AST/ALT >2xULN)
* Creatinine clearance < 30 mL/min
* Pregnant or lactating women
* Non-haematological malignancy within the past 3 years (exceptions apply - see section 6.2.2)
* Patients at a high risk of venous thromboembolism due to:
* Treatment with erythropoietic stimulating agents (e.g. erythropoietin, epoetin alpha, epoetin beta, darbepoetin alfa, methoxy polyethylene glycol-epoetin beta)
* Other risk factors not listed above and unable to receive thromboprophylaxis
* Patients with untreated osteoporosis
* Patients with uncontrolled diabetes
* Patients with a known history of glaucoma
* Any other medical or psychiatric condition likely to interfere with study participation
* Receiving treatment with an experimental drug or experimental medical device. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study. Any experimental drug treatments must be stopped at least 4 weeks before planned start of lenalidomide and dexamethasone.
* Evidence of current or past hepatitis B infection. Patient should test negative for both surface antigen (HBsAg) and hepatitis B core antibody (HBcAb)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (progression defined as development of myeloma or a new plasmacytoma outside the radiotherapy field) | 3 years from date of randomisation
  Progression free survival rate and will be analysed using Kaplan-Meier survival analysis. PSF time will be measured from date of randomisation until progression or death.

SECONDARY OUTCOMES:
Overall survival | 3 years from date of randomisation
  Time from randomisation to death of any cause will be compared between arms
Time to next treatment | At any time during the trial (up to 6 years after last patient registered)
  The time from end of radiotherapy to first date of any non-protocol treatment for plasmacytoma or myeloma will be compared between arms
Response to treatment | Approximately 1 month after Lenalidomide and Dexamethasone treatment
  The number and proportion of patients on the lenalidomide + dexamethasone arm who achieve normalisation of the SFLCr and/or the disappearance of aberrant plasma cell phenotype following Lenalidomide + Dexamethasone treatment will be documented.
Safety and toxicity of adjuvant lenalidomide + dexamethasone | During, and one month post treatment (total approximately 10 months)
  During treatment and follow up, the frequency and percentages of adverse events with a maximum severity of grade 3-5 (according to CTCAE v4.03) will be collected.
Surveillance for secondary malignancies | 5 years following treatment with lenalidomide and dexamethasone
  Second primary malignancies occurring during treatment and in the 5 years after treatment will be recorded in patients on the lenalidomide + dexamethasone arm
Treatment Compliance | 9 months from beginning of treatment
  Compliance with lenalidomide and dexamethasone treatment will be assessed using descriptive statistics. The number of reductions, delays and omissions of lenalidomide and dexamethasone will be presented as well as the median time on study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roger Owen, Principal Investigator — St James's University Hospital
Locations (13):
- United Kingdom (13):
  - Royal United Hospital, Bath
  - Blackpool Victoria Hospital, Blackpool
  - University Hospital Wales, Cardiff
  - Velindre Cancer Centre, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James University Hospital, Leeds
  - University College London Hospital, London
  - The Christie Hospital, Manchester
  - Freeman Hospital, Newcastle
  - Mount Vernon Cancer Centre, Northwood
  - Royal Preston Hospital, Preston
  - Salisbury District Hospital, Salisbury
  - Southampton General Hospital, Southampton